CLINICAL TRIAL: NCT00977106
Title: Comparative Double Blind Placebo Controlled Clinical Study on Tocilizumab Rapid Efficacy on Patients Relief in rheumatoïd Arthritis With an Inadequate Response to DMARDs or Anti TNF :TORPEDO
Brief Title: TORPEDO Study: A Study on Rapid Effect of Tocilizumab in Patients With Rheumatoid Arthritis With an Inadequate Response to Disease-Modifying Antirheumatic Drugs (DMARDs) or Anti-TNF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML22017; 2008-008309-23
Record Dates: First submitted 2009-08-18; First posted 2009-09-15 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]
- 2 (Placebo Comparator)
  Interventions: Drug: placebo
- 3 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — single iv infusion 8 mg/kg
  Arms: 1
Drug: placebo — single iv infusion
  Arms: 2
Drug: tocilizumab [RoActemra/Actemra] — iv infusion 8mg/kg every 4 weeks for 11 months
  Arms: 3

SUMMARY:
This study will assess the onset and maintenance of effect of tocilizumab on relief in patients with active moderate or severe rheumatoid arthritis who have had an inadequate response to DMARDs or anti-TNF. For the first, double-blind, part of the study patients will be randomized to receive an iv infusion of either 8mg/kg tocilizumab or placebo. After 4 weeks this will be followed by 11 months treatment with tocilizumab 8mg/kg iv infusion every 4 weeks. Methotrexate or DMARD therapy will be continued throughout study treatment. Target sample size is >100.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >/= 18 years of age
* active moderate or severe rheumatoid arthritis of <10 years duration with inadequate response to methotrexate or anti-TNF
* on methotrexate treatment for at least 10 weeks, at least 8 weeks on stable dose
* patients receiving oral corticosteroids and/or NSAIDs should be at stable dose for 4 weeks

Exclusion Criteria:

* rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA
* functional class IV by ACR classification
* history of inflammatory joint disease other than RA
* previous treatment with cell-depleting therapies, abatacept or rituximab
* active current or history of recurrent infection, or any major episode of infection requiring hospitalization or treatment with iv antibiotics <4 weeks or oral antibiotics <2 weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- France (19):
  - Amiens
  - Bayonne
  - Bois-Guillaume
  - Bordeaux
  - Brest
  - Cahors
  - Chambray-lès-Tours
  - Clermont-Ferrand
  - Échirolles
  - La Roche-sur-Yon
  - Limoges
  - Lyon
  - Metz
  - Nantes
  - Orléans
  - Paris
  - Rennes
  - Saint-Priest-en-Jarez
  - Toulouse

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Tocilizumab: Participants received placebo solution (containing polysorbate 80, sucrose, and water for injection) intravenously (IV) during the Double-Blind Treatment Period on Day 0. Starting at Week 4, participants received tocilizumab 8 milligrams per kilogram (mg/kg; 800 mg maximum) IV, once every 4 weeks up to 11 months (up to Week 44), for a maximum of 11 infusions.
- Tocilizumab: Participants received tocilizumab IV once every 4 weeks up to 12 months (up to Week 44), for a maximum of 12 infusions.
Period: Overall Study
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Started | 47 | 56 (Includes 3 participants who were randomized to placebo, but received tocilizumab.)
Completed | 37 | 45
Not Completed | 10 | 11
Not completed — Adverse Event | 5 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants who received at least 1 treatment infusion (completed or not). Three participants were randomized to the Placebo treatment group but received tocilizumab.
Groups:
- Placebo, Tocilizumab: Participants received placebo solution (containing polysorbate 80, sucrose, and water for injection) IV during the Double-Blind Treatment Period on Day 0. Starting at Week 4, participants received tocilizumab 8 mg/kg (800 mg maximum) IV, once every 4 weeks up to 11 months (up to Week 44), for a maximum of 11 infusions.
- Total: Total of all reporting groups
Arm/Group | Placebo, Tocilizumab | Tocilizumab | Total
Number analyzed (Participants) | 50 | 53 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (11.8) | 52.8 (11.6) | 52.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 77
  Male | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Significant Improvement in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 4
Description: HAQ-DI includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0 (equals)=without difficulties; 1= with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3. Relevant clinical improvement was defined as a reduction of at least 0.22 points in HAQ-DI.
Time Frame: Week 4
Population: ITT Population
Measure: Number; unit: percentage of participants
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg (800 mg maximum) IV once every 4 weeks up to 12 months (up to Week 44), for a maximum of 12 infusions.
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
percentage of participants | 42.0 | 49.1
Statistical Analysis 1: Comparison: Placebo, Tocilizumab vs Tocilizumab; Test type: Superiority or Other; p = 0.472, Chi-squared

2. Secondary Outcome: Patient Global Assessment of Disease Activity During the Double-Blind Treatment Period
Description: Participants were asked to rate their assessment of disease activity using a visual analog scale (VAS) of 0 to 100 millimeters (mm), where 0 represented no symptoms and 100 represented severe symptoms. Participants were asked to mark the line corresponding to their assessment and the distance from the left edge was measured. A negative value in change from Baseline indicates an improvement.
Time Frame: Baseline, Weeks 1 and 4
Population: ITT Population; number (n) = number of participants assessed for the specified parameter at a given visit. Changes from baseline were described for participants without missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
mm
  Baseline (n=50,53) | 58.8 (21.1) | 64.3 (17.4)
  Week 1 (n=42,42) | 49.0 (23.2) | 54.2 (20.6)
  Change at Week 1 (n=42,42) | -11.0 (19.7) | -7.4 (17.8)
  Week 4 (n=45,51) | 49.2 (24.0) | 51.1 (22.7)
  Change at Week 4 (n=45,51) | -14.3 (23.6) | -9.6 (17.4)
Statistical Analysis 1: Comparison: Placebo, Tocilizumab vs Tocilizumab; Change at Week 1; Test type: Superiority or Other; p = 0.377, Student t-test — Between-group test (equal variances)
Statistical Analysis 2: Comparison: Placebo, Tocilizumab vs Tocilizumab; Change at Week 4; Test type: Superiority or Other; p = 0.276, Student t-test; Between-group test (unequal variances)

3. Secondary Outcome: Patient Global Assessment of Disease Activity During the Open Treatment Period
Description: Participants were asked to rate their assessment of disease activity using a VAS of 0 to 100 mm, where 0 represented no symptoms and 100 represented severe symptoms. Participants were asked to mark the line corresponding to their assessment and the distance from the left edge was measured. A negative value in change from Baseline indicates an improvement.
Time Frame: Baseline, Weeks 12, 24, 36 and 48
Population: ITT Population; 3 participants were randomized to the placebo treatment group but received tocilizumab. n=number of participants assessed for the specified parameter at a given visit. Changes from baseline were described for participants without missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 47 | 56
mm
  Baseline (n=46,56) | 51.2 (22.9) | 59.4 (21.1)
  Week 12 (n=45,51) | 36.0 (23.8) | 32.7 (24.7)
  Change at Week 12 (n=44,51) | -16.2 (27.6) | -26.7 (24.2)
  Week 24 (n=438,48) | 27.4 (21.7) | 31.4 (25.9)
  Change at Week 24 (n=42,48) | -25.3 (28.5) | -27.2 (24.5)
  Week 36 (n=39,46) | 25.7 (18.1) | 28.7 (24.5)
  Change at Week 36 (n=38,46) | -24.2 (27.8) | -29.7 (25.9)
  Week 48 (n=36,45) | 25.6 (24.4) | 26.6 (23.2)
  Change at Week 48 (n=35,45) | -24.9 (28.5) | -31.7 (23.3)

4. Secondary Outcome: Physician Global Assessment of Disease Activity During the Double-Blind Treatment Period
Description: Physicians were asked to assess disease activity of the participants using a VAS of 0 to 100 mm, where 0 represented no symptoms and 100 represented severe symptoms. Physicians were asked to mark the line corresponding to their assessment and the distance from the left edge was measured. A negative value in change from Baseline indicates an improvement.
Time Frame: Baseline and Week 4
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit. Changes from baseline were described for participants without missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
mm
  Baseline (n=50,53) | 60.8 (17.2) | 58.4 (15.3)
  Week 4 (n=50,52) | 49.2 (18.1) | 44.6 (22.5)
  Change at Week 4 (n=50,52) | -11.6 (19.3) | -14.3 (20.7)
Statistical Analysis 1: Comparison: Placebo, Tocilizumab vs Tocilizumab; Change at Week 4; Test type: Superiority or Other; p = 0.502, Student t-test; Between-group test (equal variances)

5. Secondary Outcome: Physician Global Assessment of Disease Activity During the Open Treatment Period
Description: as for outcome 4
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 47 | 56
mm
  Baseline (n=47,56) | 49.3 (18.6) | 59.6 (16.3)
  Week 12 (n=44,51) | 32.9 (20.4) | 28.3 (21.7)
  Change at Week 12 (n=44,51) | -16.5 (23.9) | -30.8 (21.7)
  Week 24 (n=42,50) | 24.3 (17.0) | 24.7 (21.1)
  Change at Week 24 (n=42,50) | -27.4 (21.3) | -34.9 (21.3)
  Week 36 (n=38,46) | 22.7 (16.5) | 23.1 (20.6)
  Change at Week 36 (n=38,46) | -28.4 (20.7) | -34.9 (23.1)
  Week 48 (n=37,44) | 16.4 (15.8) | 19.3 (18.2)
  Change at Week 48 (n=37,44) | -35.0 (23.0) | -39.4 (19.7)

6. Secondary Outcome: Patient Global Assessment of Pain During the Double-Blind Treatment Period
Description: Participants were asked to rate their assessment of pain using a VAS of 0 to 100 mm, where 0 represented no pain and 100 represented intolerable pain. Participants were asked to mark the line corresponding to their assessment and the distance from the left edge was measured. A negative value in change from Baseline indicates an improvement.
Time Frame: Baseline and Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
mm
  Baseline (n=49,51) | 60.2 (20.0) | 54.6 (21.8)
  Week 4 (n=49,53) | 49.1 (24.6) | 46.4 (27.0)
  Change at Week 4 (n=49,51) | -11.1 (25.6) | -7.3 (22.8)
Statistical Analysis 1: Comparison: Placebo, Tocilizumab vs Tocilizumab; Test type: Superiority or Other; p = 0.434, t-test, 1 sided — Between placebo and TCZ groups test (Equal Variances) at week 4

7. Secondary Outcome: Patient Global Assessment of Pain During the Open Treatment Period
Description: as for outcome 6
Time Frame: Baseline and Weeks 12, 24, 36, and 48
Population: ITT Population; 3 participants were randomized to the placebo treatment group but received tocilizumab. n=number of participants assessed at a specific visit
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 47 | 56
mm
  Baseline (n=46,54) | 48.9 (24.5) | 55.1 (22.2)
  Week 12 (n=45,51) | 29.6 (23.9) | 32.8 (24.0)
  Change at Week 12 (n=44,50) | -20.3 (27.6) | -22.2 (26.2)
  Week 24 (n=43,50) | 26.2 (21.3) | 27.7 (25.2)
  Change at Week 24 (n=42,49) | -25.0 (29.2) | -25.9 (22.0)
  Week 36 (n=39,46) | 23.1 (17.2) | 25.0 (21.3)
  Change at Week 36 (n=38,45) | -25.6 (31.0) | -28.3 (27.4)
  Week 48 (n=36,45) | 22.1 (22.9) | 23.0 (20.4)
  Change at Week 48 (n=35,44) | -28.0 (29.7) | -30.4 (25.8)

8. Secondary Outcome: Synovitis Score During the Double-Blind Treatment Period Assessed Using B-Mode Ultrasound
Description: Synovitis was assessed by ultrasonography (B-mode ultrasound and Power Doppler) and scored from "0" to "3", for each of 40 joints (5 metacarpal phalangeal [MCP; left and right] joints, 5 proximal interphalangeal [PIP; left and right] joints, left and right wrists, elbows, shoulders, knees, and ankles, and 5 metatarsal phalangeal [MTP; left and right] joints); synovitis scores were calculated by adding the sum of scores for each joint for a total score ranging from 0 to 120. A score of 0 indicated no damage and a score of 120 indicated most severe damage. Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4. A negative change from baseline indicated improvement.
Time Frame: Baseline, Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
units on a scale
  Baseline (n=50,53) | 26.4 (17.2) | 25.8 (16.8)
  Week 1 (n=49,53) | 26.4 (19.1) | 25.3 (17.6)
  Change at Week 1 (n=49,53) | -0.1 (7.1) | -0.6 (7.1)
  Week 4 (n=48,52) | 26.3 (18.9) | 21.8 (15.5)
  Change at Week 4 (n=48,52) | 0.8 (7.8) | -4.4 (10.0)
Statistical Analysis 1: Comparison: Placebo, Tocilizumab vs Tocilizumab; Change at Week 1; Test type: Superiority or Other; p = 0.692, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo, Tocilizumab vs Tocilizumab; Change at Week 4; Test type: Superiority or Other; p = 0.019, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Synovitis Score During the Double-Blind Treatment Period Assessed Using Power Doppler Ultrasound
Description: Synovitis was assessed by ultrasonography (B-mode ultrasound and Power Doppler) and scored from "0" to "3", for each of 40 joints (5 MCP [left and right] joints, 5 PIP [left and right] joints, left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints); synovitis scores were calculated by adding the sum of scores for each joint for a total score ranging from 0 to 120 (higher score=more severe disease). Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4. Negative change from baseline indicated improvement.
Time Frame: Baseline, Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
units on a scale
  Baseline (n=50,53) | 10.1 (11.2) | 10.2 (11.4)
  Week 1 (n=49,53) | 9.6 (11.9) | 8.9 (12.3)
  Change at Week 1 (n=49,53) | -0.3 (3.5) | -1.4 (4.9)
  Week 4 (n=48,52) | 10.0 (13.2) | 8.4 (12.1)
  Change at Week 4 (n=48,52) | 0.8 (7.7) | -2.0 (5.1)
Statistical Analysis 1: Comparison: Placebo, Tocilizumab vs Tocilizumab; Change at Week 1; Test type: Superiority or Other; p = 0.137, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo, Tocilizumab vs Tocilizumab; Change at Week 4; Test type: Superiority or Other; p = 0.043, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Percent Change From Baseline in Synovitis Score During the Open Treatment Period Assessed Using B-Mode Ultrasound
Description: Synovitis was assessed by ultrasonography (B-mode ultrasound and Power Doppler) and scored from "0" to "3", for each of 40 joints (5 MCP [left and right] joints, 5 PIP [left and right] joints, left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints); synovitis scores were calculated by adding the sum of scores for each joint for a total score ranging from 0 to 120 (higher score=more severe disease). Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4. Relative change was the percentage (%) change from baseline.
Time Frame: Weeks 12, 24, and 48
Population: One-Year Efficacy Population: all randomized participants with at least 1 tocilizumab infusion (completed or not). n=number of participants assessed for the specified parameter at a given visit. Changes from baseline were described for participants without missing data.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo, Tocilizumab: Participants received either tocilizumab 8 mg/kg (800 mg maximum) IV or placebo solution (containing polysorbate 80, sucrose, and water for injection) IV during the Double-Blind Treatment Period on Day 0. Starting at Week 4 (Open Treatment Period), all participants received tocilizumab 8 mg/kg (800 mg maximum) IV, once every 4 weeks up to 11 months (up to Week 44), for a maximum of 11 infusions.
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 94
percent change
  Week 12 (n=94) | -15.0 (81.9)
  Week 24 (n=87) | -30.5 (64.4)
  Week 48 (n=77) | -43.7 (67.0)

11. Secondary Outcome: Percent Change From Baseline in Synovitis Score During the Open Treatment Period Assessed Using Power Doppler Ultrasound
Description: Synovitis was assessed by ultrasonography (B-mode ultrasound and Power Doppler) and scored from "0" to "3", for each of 40 joints (5 MCP [left and right] joints, 5 PIP [left and right] joints, left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints); synovitis scores were calculated by adding the sum of scores for each joint for a total score ranging from 0 to 120 (higher score=more severe disease). Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4. Relative change was the percentage change from baseline.
Time Frame: Weeks 12, 24, and 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 94
percent change
  Week 12 (n=94) | 121.0 (573.0)
  Week 24 (n=87) | -23.5 (92.8)
  Week 48 (n=77) | 3.6 (263.2)

12. Secondary Outcome: Erythrocyte Sedimentation Rate During the Double-Blind Treatment Period
Description: Erythrocyte sedimentation rate is a biological marker of inflammation, measured in mm per hour (mm/hr). A reduction in ESR indicates improvement.
Time Frame: Baseline, Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
mm/hr
  Baseline (n=50,53) | 27.5 (22.9) | 28.1 (25.6)
  Week 1 (n=49,51) | 27.6 (24.2) | 11.9 (12.7)
  Week 4 (n=50,51) | 26.6 (19.9) | 8.2 (11.0)

13. Secondary Outcome: Percent Change From Baseline in Erythrocyte Sedimentation Rate During the Double-Blind Treatment
Description: Erythrocyte sedimentation rate is a biological marker of inflammation. A negative change indicates improvement.
Time Frame: Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 49 | 53
percent change
  Week 1 (n=49,53) | 8.7 (56.4) | -51.2 (32.8)
  Week 4 (n=48,52) | 11.5 (64.1) | -65.9 (28.4)

14. Secondary Outcome: Erythrocyte Sedimentation Rate During the Open Treatment Period
Description: Erythrocyte sedimentation rate is a biological marker of inflammation, measured in mm/hr. A reduction in ESR indicates improvement. Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 103
mm/hr
  Baseline (n=103) | 27.8 (22.8)
  Week 12 (n=96) | 6.8 (11.4)
  Week 24 (n=92) | 5.9 (6.1)
  Week 36 (n=84) | 8.0 (13.4)
  Week 48 (n=80) | 4.6 (3.5)

15. Secondary Outcome: C-Reactive Protein During the Double-Blind Treatment Period
Description: C-Reactive protein (CRP) is a biological marker of inflammation and is measured in nanograms per milliliter (ng/mL). A reduction in CRP indicates improvement.
Time Frame: Baseline, Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 48 | 53
ng/mL
  Baseline (n=47,53) | 18.6 (23.6) | 14.2 (21.8)
  Week 1 (n=47,52) | 20.4 (34.3) | 2.3 (2.0)
  Week 4 (n=48,52) | 17.5 (21.8) | 3.8 (9.4)

16. Secondary Outcome: Percent Change From Baseline in C-Reactive Protein During the Double-Blind Treatment Period
Description: C-Reactive protein (CRP) is a biological marker of inflammation. Negative changes from baseline indicate improvement.
Time Frame: Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 46 | 52
percent change
  Week 1 (n=44,52) | 19.2 (70.1) | -66.2 (31.8)
  Week 4 (n=46,52) | 18.3 (95.6) | -47.0 (95.9)

17. Secondary Outcome: C- Reactive Protein During the Open Treatment Period
Description: C-reactive protein is a biological marker of inflammation and is measured in nanograms per milliliter (ng/mL). Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: ng/L
Groups:
- Placebo, Tocilzumab: Participants received either tocilizumab 8 mg/kg (800 mg maximum) IV or placebo solution (containing polysorbate 80, sucrose, and water for injection) IV during the Double-Blind Treatment Period on Day 0. Starting at Week 4 (Open Treatment Period), all participants received tocilizumab 8 mg/kg (800 mg maximum) IV, once every 4 weeks up to 11 months (up to Week 44), for a maximum of 11 infusions.
Arm/Group | Placebo, Tocilzumab
Number analyzed (Participants) | 102
ng/L
  Baseline (n=102) | 15.8 (20.8)
  Week 12 (n=95) | 3.9 (9.7)
  Week 24 (n=92) | 3.2 (5.2)
  Week 36 (n=80) | 3.9 (6.6)
  Week 48 (n=81) | 2.6 (2.6)

18. Secondary Outcome: Serum Amyloid A Component During the Double-Blind Treatment Period
Description: Serum Amyloid A (SAA) component is a biological marker of inflammation and is measured in mg/L. A reduction in SAA indicates improvement.
Time Frame: Baseline, Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 26 | 29
mg/L
  Baseline (n=23,32) | 72.0 (221.9) | 57.9 (108.2)
  Week 1 (n=26,29) | 89.5 (271.2) | 6.7 (3.6)
  Week 4 (n=25,27) | 61.2 (169.2) | 8.9 (10.4)

19. Secondary Outcome: Percent Change From Baseline in Serum Amyloid A Component During the Double-Blind Treatment Period
Description: Serum Amyloid A (SAA) component is a biological marker of inflammation. A negative change from baseline indicates improvement.
Time Frame: Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 22 | 28
percent change
  Week 1 (n=22,28) | 59.5 (247.9) | -41.2 (61.3)
  Week 4 (n=21,26) | -5.8 (39.3) | -35.5 (61.0)

20. Secondary Outcome: Serum Amyloid A Component During the Open Treatment Period
Description: Serum Amyloid A (SAA) component is a biological marker of inflammation measured in mg/L. Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo, Tocilzumab
Number analyzed (Participants) | 58
mg/L
  Baseline (n=58) | 58.6 (135.9)
  Week 12 (n=46) | 40.3 (218.7)
  Week 24 (n=46) | 13.3 (41.6)
  Week 36 (n=38) | 7.3 (6.3)
  Week 48 (n=37) | 5.7 (3.0)

21. Secondary Outcome: Beta 2 Microglobulin Levels During the Open Treatment Period
Description: Beta 2 Microglobulin is a biological marker of inflammation measured in micrograms per milliliter (mcg/mL). Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population;n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Placebo, Tocilzumab
Number analyzed (Participants) | 96
mcg/mL
  Baseline (n=96) | 2.0 (0.6)
  Week 12 (n=87) | 2.0 (0.6)
  Week 24 (n=78) | 1.9 (0.6)
  Week 36 (n=69) | 2.0 (0.5)
  Week 48 (n=64) | 1.9 (0.5)

22. Secondary Outcome: Beta 2 Microglobulin Levels During the Double-Blind Treatment Period
Description: Beta 2 Microglobulin is a biological marker of inflammation measured in micrograms per milliliter (mcg/mL).
Time Frame: Baseline, Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 45 | 49
mg/L
  Baseline (n=39,49) | 2.0 (0.6) | 2.0 (0.6)
  Week 1 (n=45,48) | 2.0 (0.5) | 2.1 (0.7)
  Week 4 (n=45,47) | 2.0 (0.5) | 2.0 (0.5)

23. Secondary Outcome: Percent Change From Baseline in Beta 2 Microglobulin Levels During the Double-Blind Treatment Period
Description: Beta 2 Microglobulin is a biological marker of inflammation. If baseline value was equal to 0, it was replaced by 0.1 to calculate the change from baseline.
Time Frame: Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 38 | 44
percent change
  Week 1 (n=38,44) | 2.2 (18.1) | 4.2 (19.6)
  Week 4 (n=37,44) | -2.3 (14.1) | -0.8 (19.4)

24. Secondary Outcome: Bone Mineral Density
Description: To describe bone mineral density (BMD), standardized values were calculated for lumbar spine, hip, femoral neck, and trochanter, taking into account the type of Dual energy X ray absorptiometry (DXA) used. All DXA at baseline were taken into account (done from before screening to Week 8). DXA at end of study were taken into account if they were done after at least 6 infusions of tocilizumab. Values were measured in milligrams per square centimeter (mg/cm^2).
Time Frame: Baseline and Week 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/cm^2
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 90
mg/cm^2
  Lumbar spine, Baseline (n=89) | 1018.0 (155.4)
  Lumbar spine, Week 48 (n=82) | 1033.4 (157.9)
  Hip, Baseline (n=90) | 887.3 (129.8)
  Hip, Week 48 (n=83) | 891.3 (131.6)
  Femoral neck, Baseline (n=90) | 825.0 (122.7)
  Femoral neck, Week 48 (n=83) | 821.8 (121.6)
  Trochanter, Baseline (n=90) | 696.2 (124.3)
  Trochanter, Week 48 (n=83) | 700.3 (122.7)

25. Secondary Outcome: Percentage of Participants Treated With Corticosteroids Over the 1-Year Tocilizumab Period
Time Frame: Baseline, Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 103
percentage of participants
  Baseline (n=103) | 74
  Week 8 (n=99) | 74
  Week 12 (n=97) | 71
  Week 16 (n=95) | 71
  Week 20 (n=93) | 70
  Week 24 (n=93) | 71
  Week 28 (n=91) | 68
  Week 32 (n=90) | 68
  Week 36 (n=85) | 69
  Week 40 (n=82) | 65
  Week 44 (n=82) | 60
  Week 48 (n=82) | 60

26. Secondary Outcome: S-Sclerostin and P-Dkk1 (Wnt Signaling Inhibitor Dickkopf) Over the 1-Year Tocilizumab Period
Description: S-Sclerostin and P-Dkk1 are biological markers of bone and cartilage metabolism measured as picograms/milliliter (pg/mL). Baseline is the closest value plus or minus (+/-) 1 month around the first tocilizumab infusion. If values before and after the first infusion were eligible, the value before was taken into account.
Time Frame: Baseline, Weeks 12, 24, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 103
pg/mL
  S-Sclerostin, Baseline (n=103) | 0.51 (0.22)
  S-Sclerostin, Week 12 (n=93) | 0.55 (0.20)
  S-Sclerostin, Week 24 (n=84) | 0.51 (0.19)
  S-Sclerostin, Week 48 (n=75) | 0.54 (0.21)
  P-Dkk1, Baseline (n=102) | 847.50 (610.22)
  P-Dkk1, Week 12 (n=86) | 572.45 (350.85)
  P-Dkk1, Week 48 (n=72) | 685.79 (482.73)

27. Secondary Outcome: Serum Procollagen Type II N-Propeptide (s-PIINP), Serum Procollagen Type I N Propeptide (s-PINP), and Serum Carboxy-Terminal Collagen Crosslinks-1 (s-CTX-I) Over the 1-Year Tocilizumab Period
Description: S-PIIINP, S-CTX-I, and S-PINP are biological markers of bone and cartilage metabolism. Baseline is the closest value +/- 1 month around the first tocilizumab infusion. If values before and after the first infusion were eligible, the value before was taken into account.
Time Frame: Baseline and Weeks 12, 24, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Tocilzumab
Number analyzed (Participants) | 103
ng/mL
  s-PIIINP, Baseline (n=103) | 5.59 (2.06)
  s-PIIINP, Week 12 (n=94) | 6.07 (2.39)
  s-PIIINP, Week 24 (n=85) | 5.74 (2.27)
  s-PIIINP, Week 48 (n=77) | 5.86 (2.12)
  s-CTX-I, Baseline (n=103) | 0.35 (0.22)
  s-CTX-I, Week 12 (n=93) | 0.35 (0.20)
  s-CTX-I, Week 48 (n=77) | 0.33 (0.18)
  s-PINP, Baseline (n=103) | 41.15 (23.95)
  s-PINP, Week 12 (n=93) | 52.33 (32.66)
  s-PINP, Week 48 (n=77) | 53.16 (30.14)

28. Secondary Outcome: Serum Osteogenic Growth Peptide (s-OGP) Over the 1-Year Tocilizumab Period
Description: S-OGP is a biological marker of bone and cartilage metabolism measured as picomoles per liter (pmol/L). Baseline is the closest value +/- 1 month around the first tocilizumab infusion. If values before and after the first infusion were eligible, the value before was taken into account.
Time Frame: Baseline and Weeks 12 and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Placebo, Tocilzumab
Number analyzed (Participants) | 103
pmol/L
  Baseline (n=103) | 3.97 (1.27)
  Week 12 (n=93) | 3.94 (1.20)
  Week 48 (n=77) | 3.90 (1.21)

29. Secondary Outcome: Weekly Methotrexate (MTX) Dose
Description: Before entering the study, participants had to be treated with MTX for at least 12 weeks and at a stable dose for at least 8 weeks before the screening visit (10-25 mg per week [mg/week] of oral or parenteral MTX). During the study, treatment with MTX had to be stable during the first month and then could be continued or modified, at the investigator's discretion.
Time Frame: Baseline and Weeks 24 and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Placebo, Tocilzumab
Number analyzed (Participants) | 103
mg/week
  Baseline (n=103) | 17.7 (4.2)
  Week 24 (n=91) | 17.1 (4.4)
  Week 48 (n=77) | 16.9 (4.6)

30. Secondary Outcome: HAQ-DI During the Double-Blind Treatment Period
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Screening and Week 4
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
units on a scale
  Screening (n=50,53) | 1.62 (0.56) | 1.60 (0.58)
  Week 4 (n=50,51) | 1.44 (0.60) | 1.39 (0.65)
  Change at Week 4 (n=50,51) | -0.18 (0.47) | -0.22 (0.49)

31. Secondary Outcome: HAQ-DI During the Open Treatment Period
Description: as for outcome 30
Time Frame: Baseline and Weeks 12, 24, 36, and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 47 | 56
units on a scale
  Baseline (n=47,56) | 1.45 (0.61) | 1.62 (0.57)
  Week 12 (n=45,49) | 1.19 (0.68) | 1.06 (0.70)
  Change at Week 12 (n=45,49) | -0.29 (0.52) | -0.62 (0.62)
  Week 24 (n=39,50) | 1.00 (0.69) | 1.01 (0.71)
  Change at Week 24 (n=39,50) | -0.50 (0.54) | -0.68 (0.61)
  Week 36 (n=39,45) | 1.05 (0.76) | 1.02 (0.71)
  Change at Week 36 (n=39,45) | -0.44 (0.75) | -0.64 (0.64)
  Week 48 (n=37,45) | 0.98 (0.78) | 0.95 (0.63)
  Change at Week 48 (n=37,45) | -0.47 (0.71) | -0.72 (0.60)

32. Secondary Outcome: Functional Assessment of Chronic Illness in Therapy - Fatigue (FACIT-F) During the Double-Blind Treatment Period
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the patient's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-F score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the participant's health status. Baseline = Last available value before Day 0 (screening or Day 0) for participants with first tocilizumab infusion at Day 0 and last value available before Week 4 (Week 1 or Week 4) for participants with first tocilizumab infusion at Week 4.
Time Frame: Day 0, Week 1, and Week 4
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
units on a scale
  Day 0 (n=50,52) | 23.9 (10.1) | 26.0 (10.6)
  Week 1 (n=48,52) | 27.3 (11.7) | 27.7 (10.4)
  Week 4 (n=49,52) | 29.2 (11.0) | 28.9 (11.0)

33. Secondary Outcome: Percent Change From Baseline in FACIT-F During the Double-Blind Treatment Period
Description: as for outcome 32
Time Frame: Week 1 and Week 4
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 49 | 52
percent change
  Week 1 (n=48,51) | 24.6 (29.0) | 22.7 (61.5)
  Week 4 (n=49,52) | 37.7 (77.1) | 41.7 (167.9)

34. Secondary Outcome: FACIT-F During the Open Treatment Period
Description: as for outcome 32
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilzumab
Number analyzed (Participants) | 102
units on a scale
  Baseline (n=102) | 27.1 (11.1)
  Week 12 (n=93) | 33.7 (11.2)
  Week 24 (n=90) | 35.4 (10.4)
  Week 36 (n=82) | 34.0 (10.3)
  Week 48 (n=82) | 34.9 (10.6)

35. Secondary Outcome: Hemoglobin Concentration During the Double-Blind Treatment Period
Description: Hemoglobin concentrations were determined at each visit to evaluate anemia in participants and measured as grams per deciliter (g/dL).
Time Frame: Baseline and Weeks 1 and 4
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
g/dL
  Baseline (n=50,53) | 12.97 (1.37) | 12.74 (1.49)
  Week 1 (n=50,51) | 12.96 (1.33) | 13.04 (1.38)
  Change at Week 1 (n=50,51) | -0.01 (0.54) | 0.34 (0.54)
  Week 4 (n=50,53) | 12.88 (1.46) | 13.10 (1.41)
  Change at Week 4 (n=50,53) | -0.09 (0.54) | 0.36 (0.69)

36. Secondary Outcome: Hemoglobin Concentration During the Open Treatment Period
Description: Hemoglobin concentrations were determined at each visit to evaluate anemia in participants and measured as g/dL.
Time Frame: Baseline, Weeks 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo, Tocilzumab
Number analyzed (Participants) | 103
g/dL
  Baseline (n=103) | 12.80 (1.47)
  Week 8 (n=99) | 13.14 (1.41)
  Week 12 (n=97) | 13.37 (1.40)
  Week 16 (n=95) | 13.24 (1.51)
  Week 20 (n=91) | 13.27 (1.46)
  Week 24 (n=92) | 13.38 (1.43)
  Week 28 (n=91) | 13.47 (1.32)
  Week 32 (n=90) | 13.46 (1.35)
  Week 36 (n=84) | 13.50 (1.31)
  Week 40 (n=81) | 13.49 (1.35)
  Week 44 (n=82) | 13.48 (1.37)
  Week 48 (n=81) | 13.64 (1.32)

37. Secondary Outcome: Tender Joint Count (TJC) Based on 28-Joint Count During the Double-Blind Treatment Period
Description: Twenty-eight joints were assessed for tenderness. Joints were classified as tender (1)/not tender (0) giving a total possible TJC score of 0 to 28. Baseline = value at Day 0 if available, value at screening otherwise.
Time Frame: Baseline and Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
tender joints
  Baseline (n=50,53) | 12.0 (6.6) | 13.4 (6.7)
  Week 1 (n=49,53) | 11.0 (7.1) | 10.6 (6.7)
  Week 4 (n=50,53) | 10.6 (6.7) | 9.9 (7.7)

38. Secondary Outcome: Percent Change From Baseline in TJC Based on 28-Joint Count During the Double-Blind Treatment Period
Description: Twenty-eight joints were assessed for tenderness. Joints were classified as tender (1)/not tender (0) giving a total possible TJC score of 0 to 28.
Time Frame: Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
percent change
  Week 1 (n=49,53) | 3.4 (74.4) | 16.7 (266.7)
  Week 4 (n=50,53) | 25.7 (180.4) | 9.3 (268.6)

39. Secondary Outcome: TJC Based on 28-Joint Count During the Open Treatment Period
Description: Twenty-eight joints were assessed for tenderness and joints were classified as tender (1)/not tender (0), giving a total possible tender joint count score of 0 to 28. Baseline = Last value available before Day 0 (selection or Day 0) for placebo and last value available before Week 4 (Week 1 or Week 4) for tocilizumab group.
Time Frame: Baseline and Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 103
tender joints
  Baseline (n=103) | 12.3 (6.9)
  Week 12 (n=97) | 5.5 (5.6)
  Week 24 (n=92) | 4.0 (4.7)
  Week 36 (n=84) | 3.6 (4.5)
  Week 48 (n=82) | 3.3 (4.7)

40. Secondary Outcome: TJC Based on 40-Joint Count During the Double-Blind Treatment Period
Description: Forty joints were assessed for tenderness (5 MCP [left and right] joints, 5 PIP [left and right joints], left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints). Joints were classified as tender (1)/not tender (0) giving a total possible TJC score of 0 to 40. Baseline = value at Day 0 if available, value at screening otherwise.
Time Frame: Baseline and Weeks 1 and 4
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit. Changes from baseline were described for participants without missing data.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
tender joints
  Baseline (n=50,53) | 17.7 (9.1) | 18.3 (8.0)
  Week 1 (n=49,53) | 16.3 (9.9) | 14.6 (9.4)
  Week 4 (n=50,53) | 15.0 (8.6) | 14.0 (10.7)

41. Secondary Outcome: Percent Change From Baseline in TJC Based on 40-Joint Count During the Double-Blind Treatment Period
Description: Forty joints were assessed for tenderness (5 MCP [left and right] joints, 5 PIP [left and right joints], left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints). Joints were classified as tender (1)/not tender (0) giving a total possible TJC score of 0 to 40.
Time Frame: Weeks 1 and 4
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
percent change
  Week 1 (n=49,53) | -2.6 (59.5) | -22.1 (39.6)
  Week 4 (n=50,53) | -1.5 (63.5) | -23.1 (49.3)

42. Secondary Outcome: TJC Based on 40-Joint Count During the Open Treatment Period
Description: Forty joints were assessed for tenderness (5 MCP [left and right] joints, 5 PIP [left and right joints], left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints). Joints were classified as tender (1)/not tender (0) giving a total possible TJC score of 0 to 40. Baseline = Last value available before Day 0 (selection or Day 0) for placebo and last value available before Week 4 (Week 1 or Week 4) for tocilizumab group.
Time Frame: Baseline and Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 103
tender joints
  Baseline (n=103) | 17.0 (8.7)
  Week 12 (n=97) | 7.9 (7.7)
  Week 24 (n=92) | 5.9 (6.5)
  Week 36 (n=84) | 5.2 (6.2)
  Week 48 (n=82) | 5.0 (6.5)

43. Secondary Outcome: Swollen Joint Count (SJC) Based on 28-Joint Count During the Double-Blind Treatment Period
Description: Twenty-eight joints were assessed for swelling. Joints were classified as swollen (1)/not swollen (0) giving a total possible SJC score of 0 to 28. Baseline = value at Day 0 if available, value at screening otherwise.
Time Frame: Baseline and Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
swollen joints
  Baseline (n=50,53) | 8.3 (4.2) | 8.5 (4.5)
  Week 1 (n=49,53) | 6.9 (4.4) | 7.0 (4.8)
  Week 4 (n=50,53) | 7.7 (4.6) | 5.8 (3.8)

44. Secondary Outcome: Percent Change From Baseline in SJC Based on 28-Joint Count During the Double-Blind Treatment Period
Description: Twenty-eight joints were assessed for swelling. Joints were classified as swollen (1)/not swollen (0) giving a total possible SJC score of 0 to 28.
Time Frame: Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
percent change
  Week 1 (n=49,53) | -12.0 (54.0) | -10.9 (70.6)
  Week 4 (n=50,53) | -1.1 (53.7) | -27.3 (47.6)

45. Secondary Outcome: Swollen Joint Count (SJC) Based on 28-Joint Count During the Open Treatment Period
Description: Twenty-eight joints were assessed for swelling (5 MCP [left and right] joints, 5 PIP [left and right joints], left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints) . Joints were classified as swollen (1)/not swollen (0) giving a total possible SJC score of 0 to 28. Baseline = Last value available before Day 0 (selection or Day 0) for placebo and last value available before Week 4 (Week 1 or Week 4) for tocilizumab group.
Time Frame: Baseline and Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 103
swollen joints
  Baseline (n=103) | 8.2 (4.6)
  Week 12 (n=97) | 3.8 (4.0)
  Week 24 (n=92) | 3.1 (3.4)
  Week 36 (n=84) | 2.2 (3.0)
  Week 48 (n=82) | 1.7 (2.6)

46. Secondary Outcome: SJC Based on 40-Joint Count During the Double-Blind Treatment Period
Description: Forty joints were assessed for swelling (5 MCP [left and right] joints, 5 PIP [left and right joints], left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints). Joints were classified as swollen (1)/not swollen (0) giving a total possible SJC score of 0 to 40. Baseline = value at Day 0 if available, value at screening otherwise.
Time Frame: Baseline and Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
swollen joints
  Baseline (n=50,53) | 10.1 (5.0) | 10.4 (5.1)
  Week 1 (n=49,53) | 8.7 (5.3) | 8.0 (5.3)
  Week 4 (n=50,53) | 9.8 (6.0) | 6.7 (4.5)

47. Secondary Outcome: Percent Change From Baseline in SJC Based on 40-Joint Count During the Double-Blind Treatment Period
Description: Forty joints were assessed for swelling (5 MCP [left and right] joints, 5 PIP [left and right joints], left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints). Joints were classified as swollen (1)/not swollen (0) giving a total possible SJC score of 0 to 40.
Time Frame: Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
percent change
  Week 1 (n=49,53) | -9.2 (58.1) | -19.2 (45.3)
  Week 4 (n=50,53) | 7.7 (73.8) | -30.0 (45.9)

48. Secondary Outcome: SJC Based on 40-Joint Count During the Open Treatment Period
Description: Forty joints were assessed for swelling (5 MCP [left and right] joints, 5 PIP [left and right joints], left and right wrists, elbows, shoulders, knees, and ankles, and 5 MTP [left and right] joints). Joints were classified as swollen (1)/not swollen (0) for a total possible score of 0 to 40. Baseline = Last value available before Day 0 (selection or Day 0) for placebo and last value available before Week 4 (Week 1 or Week 4) for tocilizumab group.
Time Frame: Baseline and Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 103
swollen joints
  Baseline (n=103) | 10.2 (5.7)
  Week 12 (n=97) | 4.4 (4.7)
  Week 24 (n=92) | 3.5 (3.7)
  Week 36 (n=84) | 2.5 (3.3)
  Week 48 (n=82) | 2.1 (3.0)

49. Secondary Outcome: Disease Activity Score Based on 28-Joints Count (DAS28) During the Double-Blind Treatment Period
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, the erythrocyte sedimentation rate and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 less than or equal to (≤3.2) = low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
units on a scale
  Baseline (n=50,53) | 5.66 (1.02) | 5.64 (1.04)
  Week 1 (n=41,40) | 5.40 (1.04) | 4.41 (1.05)
  Change at Week 1 (n=41,40) | -0.43 (0.81) | -1.12 (0.61)
  Week 4 (n=45,50) | 5.27 (1.00) | 4.00 (1.26)
  Change at Week 4 (n=45,50) | -0.43 (0.90) | -1.68 (0.94)

50. Secondary Outcome: DAS28 During the Open Treatment Period
Description: as for outcome 49
Time Frame: Baseline and Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 103
units on a scale
  Baseline (n=102) | 5.51 (1.04)
  Week 12 (n=95) | 2.98 (1.40)
  Week 24 (n=89) | 2.64 (1.31)
  Week 36 (n=83) | 2.51 (1.36)
  Week 48 (n=79) | 2.22 (1.28)

51. Secondary Outcome: Disease Activity Score Based on 40-Joints Count (DAS40) During the Double-Blind Treatment Period
Description: DAS40 calculated from the number of swollen joints and tender joints using the 40-joint count, the erythrocyte sedimentation rate and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity.
Time Frame: Baseline and Weeks 1 and 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab | Tocilizumab
Number analyzed (Participants) | 50 | 53
units on a scale
  Baseline (n=50,53) | 6.15 (1.03) | 6.08 (1.04)
  Week 1 (n=41,40) | 5.88 (1.12) | 4.71 (1.16)
  Change at Week 1 (n=41,40) | -0.43 (0.85) | -1.25 (0.64)
  Week 4 (n=45,50) | 5.70 (1.03) | 4.39 (1.37)
  Change at Week 4 (n=45,50) | -0.49 (1.03) | -1.75 (1.03)

52. Secondary Outcome: DAS40 During the Open Treatment Period
Description: DAS40 was calculated from the number of swollen joints and tender joints using the 40-joint count, the erythrocyte sedimentation rate, and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS40 score ranged from 0 to 10, where higher scores correspond to greater disease activity.
Time Frame: Baseline and Weeks 12, 24, 36, and 48
Population: One-Year Efficacy Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Tocilizumab
Number analyzed (Participants) | 102
units on a scale
  Baseline (n=102) | 5.96 (1.06)
  Week 12 (n=95) | 3.27 (1.49)
  Week 24 (n=89) | 2.89 (1.40)
  Week 36 (n=83) | 2.76 (1.42)
  Week 48 (n=79) | 2.48 (1.40)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the study, from date of Screening until the end of study at Week 48.
Arm/Group | Tocilizumab | Placebo, Tocilizumab
Serious Adverse Events (participants affected / at risk) | 13/53 | 11/50
Other Adverse Events (participants affected / at risk) | 30/53 | 15/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=53) | Placebo, Tocilizumab (N=50)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
ALT increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=53) | Placebo, Tocilizumab (N=50)
Bronchitis (Infections and infestations) | 7 | 8
Gastroenteritis (Infections and infestations) | 9 | 4
Influenza (Infections and infestations) | 3 | 2
Oral herpes (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 7 | 3
Folliculitis (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 4 | 1
Rhinitis (Infections and infestations) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4
Aphthous stomatitis (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 3 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 7 | 4
Burning sensation (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 4 | 3
Presyncope (Nervous system disorders) | 4 | 0
Sciatica (Nervous system disorders) | 3 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 6
Asthenia (General disorders) | 6 | 3
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 2 | 0
Weight increased (Investigations) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 3 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 2 | 0
Stress (Psychiatric disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 0
Auricular pseudocyst (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 10 | 7
Tonsillitis (Infections and infestations) | 4 | 3
Sinusitis (Infections and infestations) | 2 | 3
Herpes zoster (Infections and infestations) | 1 | 2
Escherichia urinary tract infection (Infections and infestations) | 2 | 0
Laryngitis (Infections and infestations) | 2 | 0
Oral fungal infection (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 2
Bacterial infection (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Dermo-hypodermitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1
Nail bed infection (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Vaginitis gardnerella (Infections and infestations) | 1 | 0
Viral tonsillitis (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Transaminases increased (Investigations) | 2 | 3
Hepatic enzyme increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast discomfort (Reproductive system and breast disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Cerumen removal (Surgical and medical procedures) | 1 | 0
Gingival operation (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0
Thalassaemia beta (Congenital, familial and genetic disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 4
Biliary cyst (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Xerophthalmia (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 1
Chalazion (Eye disorders) | 1 | 0
Eyelid cyst (Eye disorders) | 0 | 2
Conjunctivitis (Eye disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Gingival recession (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Aerophagia (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Tooth discolouration (Gastrointestinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotrichosis (Skin and subcutaneous tissue disorders) | 0 | 1
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Fatigue (General disorders) | 2 | 3
Chest discomfort (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Site of oppression (General disorders) | 1 | 0
Vaccination site haematoma (General disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Vascular disorders) | 1 | 4
Hot flush (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous insufficiency (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.